CLINICAL TRIAL: NCT02193815
Title: A Phase 1, Single- Center, Randomized, Double-blind, Vehicle And Active Comparator-controlled Trial To Evaluate The Antipsoriatic Activity And Safety Of A Topically Applied Pf-06263276 Formulation In A Psoriasis Plaque Test
Brief Title: A 12 Day Study To Evaluate A Topical Drug To Treat Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B5391003; 2014-000068-16 (EudraCT Number)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Psoriasis Vulgaris
Keywords: psoriasis; plaque; vulgaris; phase 1; randomized; double-blind; topical; safety
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid | interventions — PF-06263276; calcipotriene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- One Arm (Experimental): Study treatments 1-6 Study drug, vehicle, Tofacitinib, vehicle, Daivonex solution and ointment
  Interventions: Drug: PF06263276; Other: Vehicle; Drug: 2%Tofacitinib Ointment; Drug: Daivonex; Drug: Daivonex Ointment

INTERVENTIONS:
Drug: PF06263276 — 4% PF 06263276 solution Daily dosage: approximately 8 mg PF 06263276 QD
Other: Vehicle — Active ingredient-free vehicle to 4% solution
Drug: 2%Tofacitinib Ointment — Daily Dosage: approximately 4 mg tofacitinib
Other: Vehicle — Active ingredient-free vehicle to 2% Ointment
Drug: Daivonex — Daivonex solution (50 ug/ml Calcipotriol) Daily Dosage of calcipotriol: approximately 0.01 mg
Drug: Daivonex Ointment — Daivonex ointment (50 ug/g Calcipotriol) Daily Dosage of calcipotriol: approximately 0.01 mg

SUMMARY:
This is a vehicle and comparator controlled Proof of Mechanism (PoM) trial to evaluate the effect on psoriasis disease activity and safety of topically applied PF 06263276 in subjects with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects age 18 years and older, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.
* Subjects with psoriasis vulgaris in a chronic stable phase and with a plaque area of mild to moderate severity sufficient for six treatment fields located in up to three plaque areas.
* The target lesion(s) should be on the trunk or extremities (excluding palms/soles). Psoriatic lesions on the knees or elbows are not to be used as a target lesion.

Exclusion Criteria:

* Subjects with psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica, psoriasis arthropathica and pustular psoriasis.
* Treatment with any systemic medications which in the opinion of the investigator might counter or influence the trial aim (including anti psoriasis medications, eg, corticosteroids, cytostatics or retinoids) or medications which are known to provoke or aggravate psoriasis (eg, beta blocker, anti malarial drugs, lithium) or phototherapy/psoralen+UVA (PUVA) within 4 weeks preceding the treatment phase of the trial and during the trial.
* Treatment with any locally acting medications (including anti-psoriasis medications like vitamin D analogues, dithranol) within 4 weeks of the treatment phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Bioskin GmbH, Hamburg, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5391003&StudyName=A%2012%20Day%20Study%20To%20Evaluate%20A%20Topical%20Drug%20To%20Treat%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial enrolled participants with chronic plaque type psoriasis and with a treatment area sufficient for 6 treatment fields on 1 to 3 comparable plaques defined as having treatment fields with psoriatic skin thickness/Echo-Poor Band (EPB) of at least 200 micrometers.
Groups:
- All Participants: Participants received the following treatments topically to 6 selected treatment fields: 4% PF-06263276 and its corresponding vehicle, 2% tofacitinib and its corresponding vehicle, calcipotriol (Daivonex) solution, and Daivonex ointment. The fields were occluded and participants returned daily to the center for re-application during the 11-day treatment period.
Period: Overall Study
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who received at least 1 dose of investigational product.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriatic Skin Thickness/Echo-Poor Band (EPB) for PF-06263276 4% Solution in Comparison to Corresponding Vehicle at Day 12
Description: Psoriatic skin thickness was measured using a 20 megahertz (MHz) high frequency sonograph. Serial A-scans were composed and presented on a monitor as a section of the skin.
Time Frame: Day 1 (Baseline), Day 12
Population: The Intent-to-Treat (ITT) population included all participants who had investigational products dispensed and had at least 1 post-baseline assessment of the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: micrometers
Groups:
- PF-06263276 4% Solution: All participants who received PF-06263276 4% solution topically once daily for 11 days.
- PF-06263276 Vehicle: All participants who received PF-06263276 vehicle (active ingredient- free) topically once daily for 11 days.
Arm/Group | PF-06263276 4% Solution | PF-06263276 Vehicle
Number analyzed (Participants) | 15 | 15
micrometers
  Baseline | 358.9 (132.84) [285 to 432] | 353.1 (121.03) [286 to 420]
  Change at Day 12 | 17.7 (91.10) [-33 to 68] | 32.9 (96.72) [-21 to 86]
Statistical Analysis 1: Comparison: PF-06263276 4% Solution vs PF-06263276 Vehicle; Test type: Superiority or Other; p = 0.3465, Mixed Models Analysis; Adjusted Mean Ratio = 93.20, 95% CI 2-sided [80.43 to 107.99], Standard Error of Mean 0.075

2. Secondary Outcome: Change From Baseline in Psoriatic Skin Thickness/EPB for PF-06263276 4% Solution in Comparison to Daivonex Solution at Day 12
Time Frame: Day 1 (Baseline), Day 12
Population: The ITT population included all participants who had investigational products dispensed and had at least 1 post-baseline assessment of the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: micrometers
Groups:
- Daivonex Solution: All participants who received calcipotriol solution (50 micrograms per milliliter [mcg/mL]) topically once daily for 11 days.
Arm/Group | PF-06263276 4% Solution | Daivonex Solution
Number analyzed (Participants) | 15 | 15
micrometers | 17.7 (91.10) | -135.5 (114.27)
Statistical Analysis 1: Comparison: PF-06263276 4% Solution vs Daivonex Solution; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean = 165.88, 95% CI 2-sided [143.12 to 192.25], Standard Error of Mean 0.075

3. Secondary Outcome: Change From Baseline in Psoriatic Skin Thickness/EPB for Tofacitinib 2% Ointment in Comparison to Corresponding Vehicle at Day 12
Time Frame: Day 1 (Baseline), Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometers
Groups:
- Tofacitinib 2% Ointment: All participants who received tofacitinib 2% ointment topically once daily for 11 days.
- Tofacitinib Vehicle: All participants who received tofacitinib vehicle (active ingredient-free) topically once daily for 11 days.
Arm/Group | Tofacitinib 2% Ointment | Tofacitinib Vehicle
Number analyzed (Participants) | 15 | 15
micrometers
  Baseline | 364.1 (135.82) | 357.3 (135.60)
  Change at Day 12 | -117.8 (115.15) | 0.1 (95.04)
Statistical Analysis 1: Comparison: Tofacitinib 2% Ointment vs Tofacitinib Vehicle; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean = 65.42, 95% CI 2-sided [56.46 to 75.81], Standard Error of Mean 0.075

4. Secondary Outcome: Change From Baseline in Psoriatic Skin Thickness/EPB at Day 8
Time Frame: Day 1 (Baseline), Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometers
Groups:
- PF-06263276 Vehicle: All participants who received PF-06263276 vehicle (active ingredient-free) topically once daily for 11 days.
- Daivonex Ointment: All participants who received calcipotriol ointment (50 micrograms per gram [mcg/g]) topically once daily for 11 days.
Arm/Group | PF-06263276 4% Solution | PF-06263276 Vehicle | Tofacitinib 2% Ointment | Tofacitinib Vehicle | Daivonex Solution | Daivonex Ointment
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
micrometers
  Baseline | 358.9 (132.84) | 353.1 (121.03) | 364.1 (135.82) | 357.3 (135.60) | 376.1 (148.44) | 364.1 (124.35)
  Change at Day 8 | 18.0 (86.37) | 38.5 (65.45) | -90.5 (84.11) | 15.1 (104.55) | -98.8 (127.18) | -104.7 (65.83)
Statistical Analysis 1: Comparison: PF-06263276 4% Solution vs PF-06263276 Vehicle; Test type: Superiority or Other; p = 0.3349, Mixed Models Analysis; Adjusted Mean = 93.04, 95% CI 2-sided [80.30 to 107.81], Standard Error of Mean 0.075
Statistical Analysis 2: Comparison: PF-06263276 4% Solution vs Daivonex Solution; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean = 149.56, 95% CI 2-sided [129.04 to 173.34], Standard Error of Mean 0.075
Statistical Analysis 3: Comparison: Tofacitinib 2% Ointment vs Daivonex Ointment; Test type: Superiority or Other; p = 0.3991, Mixed Models Analysis; Adjusted Mean = 106.51, 95% CI 2-sided [91.92 to 123.41], Standard Error of Mean 0.075
Statistical Analysis 4: Comparison: Tofacitinib 2% Ointment vs Tofacitinib Vehicle; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean = 71.94, 95% CI 2-sided [62.08 to 83.36], Standard Error of Mean 0.075

5. Secondary Outcome: Area Under the Curve (AUC) of Psoriatic Skin Thickness/EPB
Description: The AUC of psoriatic skin thickness/EPB from Day 1 to Day 12 was determined using the linear trapezoidal rule. The mean raw values are reported.
Time Frame: Day 1 (baseline) up to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometers*day
Arm/Group | PF-06263276 4% Solution | PF-06263276 Vehicle | Tofacitinib 2% Ointment | Tofacitinib Vehicle | Daivonex Solution | Daivonex Ointment
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
micrometers*day | 4082.60 (1726.167) | 4161.40 (1436.733) | 3271.93 (1210.138) | 4013.07 (1465.339) | 3322.40 (1663.668) | 3165.47 (1113.937)
Statistical Analysis 1: Comparison: PF-06263276 4% Solution vs PF-06263276 Vehicle; Test type: Superiority or Other; p = 0.7529, Mixed Models Analysis; Adjusted Mean = 96.04, 95% CI 2-sided [74.00 to 124.64], Standard Error of Mean 0.127
Statistical Analysis 2: Comparison: PF-06263276 4% Solution vs Daivonex Solution; Test type: Superiority or Other; p = 0.1318, Mixed Models Analysis; Adjusted Mean = 125.62, 95% CI 2-sided [92.96 to 169.75], Standard Error of Mean 0.147
Statistical Analysis 3: Comparison: Tofacitinib 2% Ointment vs Daivonex Ointment; Test type: Superiority or Other; p = 0.8009, Mixed Models Analysis; Adjusted Mean = 103.35, 95% CI 2-sided [79.30 to 134.68], Standard Error of Mean 0.129
Statistical Analysis 4: Comparison: Tofacitinib 2% Ointment vs Tofacitinib Vehicle; Test type: Superiority or Other; p = 0.1012, Mixed Models Analysis; Adjusted Mean = 81.09, 95% CI 2-sided [62.94 to 104.47], Standard Error of Mean 0.124

6. Secondary Outcome: Global Clinical Assessment at Day 1, 8 and 12
Description: Global Clinical Assessment of the test fields was performed by visual examination using a 5-point score (-1=worsened; 0=unchanged [no effect]; 1=slight improvement; 2=clear improvement but not completely healed; 3=completely healed). Clinically apparent differences in erythema and infiltration will contribute to this global assessment. At baseline (Day 1), the score was documented as "0" (unchanged).
Time Frame: Day 1, Day 8, Day 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | PF-06263276 4% Solution | PF-06263276 Vehicle | Tofacitinib 2% Ointment | Tofacitinib Vehicle | Daivonex Solution | Daivonex Ointment
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
participants
  Day 1: Score -1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1: Score 0 | 15 | 15 | 15 | 15 | 15 | 15
  Day 1: Score 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1: Score 2 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1: Score 3 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: Score -1 | 0 | 0 | 0 | 0 | 1 | 0
  Day 8: Score 0 | 13 | 15 | 4 | 14 | 1 | 1
  Day 8: Score 1 | 2 | 0 | 8 | 0 | 9 | 6
  Day 8: Score 2 | 0 | 0 | 3 | 1 | 4 | 8
  Day 8: Score 3 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12: Score -1 | 0 | 0 | 0 | 0 | 1 | 1
  Day 12: Score 0 | 13 | 15 | 4 | 11 | 1 | 2
  Day 12: Score 1 | 2 | 0 | 8 | 3 | 6 | 4
  Day 12: Score 2 | 0 | 0 | 3 | 1 | 7 | 8
  Day 12: Score 3 | 0 | 0 | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Specified Skin AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs. The number of participants with specified skin AEs was reported.
Time Frame: Baseline up to 28 days after last study drug administration (Day 21)
Population: The safety population included all enrolled participants who received at least 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | PF-06263276 4% Solution | PF-06263276 Vehicle | Tofacitinib 2% Ointment | Tofacitinib Vehicle | Daivonex Solution | Daivonex Ointment
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
participants
  Specified Skin AEs | 0 | 0 | 0 | 0 | 0 | 2
  Specified Skin SAEs | 0 | 0 | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, RBC morphology, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (e.g., urine human chorionic gonadotropin [hCG] for females of childbearing potential).
Time Frame: Baseline up to Day 12
Population: The safety population included all enrolled participants who received at least 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
participants | 6

9. Other Pre Specified Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate <40 or >120 beats per minute (bpm), standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) >=30 millimeters of mercury (mmHg) change from baseline in same posture or SBP <90 mmHg, diastolic blood pressure (DBP) >=20 mmHg change from baseline in same posture or DBP <50 mmHg.
Time Frame: Baseline up to Day 12
Population: The safety population included all enrolled participants who received at least 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
participants
  SBP <90 mmHg | 0
  DBP <50 mmHg | 0
  Pulse Rate <40 or >120 bpm | 0
  Maximum Increase from Baseline in SBP >=30 mmHg | 0
  Maximum Increase from Baseline in DBP >=20 mmHg | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration (Day 21)
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=15)
Nausea (Gastrointestinal disorders) | 1
Facial pain (General disorders) | 1
Dizziness (Nervous system disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.